CLINICAL TRIAL: NCT00800475
Title: A Relative Bioequivalence Study of 600 mg Gemfibrozil Tablets Under Fasting Conditions
Brief Title: Bioequivalence Study Between Two Oral Formulations of Gemfibrozil Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Blu Caribe (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R05-0116
Record Dates: First submitted 2008-11-26; First posted 2008-12-02 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Bioavailability
Keywords: bioavailability; Gemfibrozil
MeSH Terms: interventions — Gemfibrozil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Drug (Active Comparator)
  Interventions: Drug: Gemfibrozil Tablets
- Reference Drug (Active Comparator)
  Interventions: Drug: Gemfibrozil Tablets

INTERVENTIONS:
Drug: Gemfibrozil Tablets

SUMMARY:
The purpose of this study is to determine whether two oral formulations of Gemfibrozil Tablets are bioequivalent.

ELIGIBILITY:
Inclusion Criteria:

* healthy men or women 18 years of age or older
* weight within +/- 20% for height and body frame
* willing to participate and sign a copy of the informed consent form

Exclusion Criteria:

* recent history of drug or alcohol addiction or abuse
* pregnant or lactating women
* history of allergic response to gemfibrozil
* use of tobacco products
* evidence of a clinically significant disorder or whose laboratory results were deemed to be clinically significant
* receipt of any drugs as part of a research study within 28 days prior to study dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-07; Primary Completion 2005-07 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalence was assessed on the pharmacokinetic variables, Cmax, AUCO-t and AUCO-infinity